CLINICAL TRIAL: NCT01895699
Title: The Effect of Contrast Agent on Endothelial Function in Healthy Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinol and Metab, Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2013Wze033
Record Dates: First submitted 2013-07-04; First posted 2013-07-10 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Contrast Agent; Endothelial Function; Cytokines; Apoptosis of Endothelial Progenitor Cell; Free Radical; Alpha-lipoic Acid
Keywords: Contrast agent; endothelium; Free radical; Alpha lipoic acid
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- contrast group (Ioversol) (Experimental): Each individual will be given 80 ml Ioversol via intravenous injection within 5 minutes
  Interventions: Other: Contrast agent
- Placebo group (Placebo Comparator)
- alpha-lipoic acid group (Other): Alpha-lipoic acid 600 mg in 0.9% sodium chloride 250 ml was administrated 1 hour before contrast agents via venous. and only 0.9% sodium chloride 250 ml was administrated for other 2 groups.
  Interventions: Other: Contrast agent

INTERVENTIONS:
Other: Contrast agent
  Arms: alpha-lipoic acid group; contrast group (Ioversol)

SUMMARY:
Contrast medium is essential for diagnosis of many diseases. However, recent studies showed that contrast agents can induce renal injury and is associated with poor long-term clinical outcome, especially in diabetes. To date, no data are available on the relationship between contrast medium and endothelial function. Endothelial dysfunction is known to precede atherosclerosis and is considered a risk marker for future development of cardiovascular disease. Therefore, we hypothesized that contrast agents may induce endothelial dysfunction in healthy men. In addition, we hypothesized that contrast induced endothelial dysfunction via free radicals. Thus, we also test alpha-lipoic acid whether or not protect endothelial dysfunction induced by contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* 20 yr < = age < = 30 yr
* 20 < = body mass index < = 25

Exclusion Criteria:

* age < 20 yr or > 30 yr
* dysfunction for liver, renal, and heart.
* other diseases such as diabetes, hypertension, thyroid disease

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The endothelial dysfunction and the protective role of alpha-lipoic acid | 6 months

SECONDARY OUTCOMES:
The apoptosis of endothelial progenitor cell | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China